CLINICAL TRIAL: NCT00701675
Title: Pharmacological Treatment of Generalized Anxiety Disorder in the Elderly
Acronym: Sert-GAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-005-04F
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: sertraline; pharmacotherapy; geriatric
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sertraline 50mg (Experimental): sertraline 50 mg daily
  Interventions: Drug: sertraline 50 mg daily
- Sertraline 100mg (Experimental): sertraline 100mg daily
  Interventions: Drug: sertraline 100 mg daily
- Placebo (Placebo Comparator): placebo 50 or 100mg
  Interventions: Drug: Placebo 50 or 100 mg

INTERVENTIONS:
Drug: sertraline 50 mg daily — 50 mg daily
  Other Names: zoloft 50 mg daily
  Arms: Sertraline 50mg
Drug: sertraline 100 mg daily — 100 mg daily
  Other Names: zoloft 100mg daily
  Arms: Sertraline 100mg
Drug: Placebo 50 or 100 mg — 50mg or 100mg matching placebo
  Other Names: 50mg or 100mg matching placebo
  Arms: Placebo

SUMMARY:
Generalized anxiety disorder (GAD) is a very common disorder in the geriatric population with prevalence rates reaching 7% and even higher rates of 8% among elderly veterans. However, despite such high prevalence treating clinicians are presently forced to address treatment issues in this population without the guidance of scientific data. This proposal aims to begin to address this void.

In light of emerging information regarding efficacy of the newer anti anxiety agents, specifically the selective serotonin reuptake inhibitors (SSRIs), in the treatment of young adult GAD patients it is time to prospectively evaluate the safety and efficacy of these medications in the treatment of elderly GAD patients. Therefore, this study will examine the effects and safety of the SSRI sertraline at different doses (50mg and 100mg per day) for older patients with GAD.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a serious and distinct illness that occurs in significant numbers, affecting at least 7 million people in the United States alone. The prevalence of GAD is higher in the primary care setting with rates twice as high as the rates reported in community samples. GAD is a life-long disorder with low remission rates, resulting in high disability and morbidity. Of significance are emerging epidemiological data suggesting that GAD is highly prevalent in the geriatric population with prevalence rates ranging from 1.9% to 7.1% and accounting for the majority of anxiety disorder cases in this age group. More alarming is the fact that the presence of anxiety symptoms leads to considerable functional impairment, increased morbidity, and mortality among the affected elderly population, thus leading to increases in the costs of their care. However, despite advances made in GAD treatment in the adult population, no prospective data are presently available on the treatment of GAD in the elderly population, forcing clinicians to provide treatment without the guidance of scientific data. These findings are of particular relevance to the Veterans Affairs Health Care System where the average age of patients treated in primary care clinics is currently 60-64 years. The present application focuses on this target subpopulation of elderly veterans.

This proposal aims to provide evidence-based guidelines for pharmacological management of elderly veterans suffering from generalized anxiety disorder. This will be accomplished by conducting a clinical trial in elderly veterans suffering from GAD by evaluating the efficacy and safety of sertraline - a proven anxiolytic compound widely used in the young adult population.

We believe that this proposed study will be one of the first studies in this area. Thus, it may also serve as a first step in a future line of research aimed at developing comprehensive pharmacological and psychosocial interventions in the treatment of anxiety in the elderly.

(b) HYPOTHESIS/RESEARCH QUESTIONS Study Hypothesis In a double-blind, placebo-controlled trial in elderly veterans diagnosed with GAD, sertraline will be more effective and equally safe as placebo in reducing symptoms of generalized anxiety disorder.

Research Question Will the presence of differences in pharmacokinetics (PK) (i.e., mean population values of steady state plasma concentrations) and plasma levels of sertraline explain differences in efficacy and side effect profile between and within the two fixed sertraline doses studied, if detected? (c) SPECIFIC OBJECTIVE The objective of the proposed study is to conduct a multi-site, double-blind, placebo-controlled trial evaluating the efficacy and safety of sertraline at fixed doses vs. placebo in the treatment of GAD among elderly primary care outpatient veterans.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race, ages 60 years and older.
* Willingness to accept randomization.
* Subjects who meet current (Diagnostic and Statistical Manual of Psychiatric Disorders forth edition (DSM-IV) criteria for a principal diagnosis of GAD
* Patients must have a minimum of a "moderately ill" rating on the Clinicians Global Impression-Severity Scale for GAD.
* Patients will have a score of 10 or more on the Hospital Anxiety and Depression Rating Scale (HADS) Anxiety subscale.
* Subjects entering the study will be free of psychotropic medications.

Exclusion Criteria:

* Subjects with DSM-IV current major depressive episode will be excluded.
* Subjects who exhibit suicidal ideation or are judged to be a significant suicide risk.
* Subjects who meet DSM-IV criteria for a substance (drug and alcohol) abuse and dependence disorder within the past 6 months
* Subjects who meet current or past DSM-IV criteria for psychotic disorder, or bipolar disorder.
* Subjects who meet DSM-IV criteria for dementia.
* Subjects with DSM-IV current major depressive episode will be excluded.
* Subjects who exhibit suicidal ideation or are judged to be a significant suicide risk.
* Subjects who meet DSM-IV criteria for a substance (drug and alcohol) abuse and dependence disorder within the past 6 months
* Subjects who meet current or past DSM-IV criteria for psychotic disorder, or bipolar disorder.
* Subjects who meet DSM-IV criteria for dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Brawman-Mintzer, MD, Principal Investigator — Ralph H Johnson VA Medical Center, Charleston
Locations (3):
- United States (3):
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline 50mg: sertraline 50mg per day
  sertraline 50 mg daily: 50 mg daily
- Sertraline 100mg: sertraline 100mg per day
  sertraline 100 mg daily: 100 mg daily
- Placebo: matching placebo
  Placebo 50 or 100 mg: matching placebo
Period: Overall Study
Arm/Group | Sertraline 50mg | Sertraline 100mg | Placebo
Started | 14 | 14 | 14
Completed | 10 | 6 | 7
Not Completed | 4 | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline 50mg | Sertraline 100mg | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 9 | 26
  >=65 years | 6 | 5 | 5 | 16
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 13 | 14 | 14 | 41
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Comparisons of End of Study HAM-A Score Means for Sertraline 50 mg vs Placebo, Sertraline 100 mg vs Placebo, and Sertraline 50 mg vs. Sertraline 100 mg
Description: Least squares (LS) means estimate and p-value from mixed effects model with baseline and site as covariates and Tukey-Kramer adjustment for multiple comparisons Hamilton Rating Scale for Anxiety (HAM-A) is a widely used rating scale for anxiety describes the presence/absence of the severity of anxiety symptoms. It's clinician-rated scale of 14 items rated from 0-4. Generally, total score of <17 is mild anxiety; 18-24 is mild to moderate, and 25 and up is moderate to severe.
Time Frame: 11 weeks from baseline
Population: sertraline 50mg group and placebo group each had 2 subjects with missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sertraline 50mg | Sertraline 100mg | Placebo
Number analyzed (Participants) | 14 | 12 | 12
units on a scale | 10.638 [7.456 to 13.819] | 10.008 [5.692 to 14.323] | 9.357 [5.159 to 13.554]

ADVERSE EVENTS:
Time Frame: weeks 1,2,3,5,7,9,and 11
Arm/Group | Sertraline 50mg | Sertraline 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 4/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline 50mg (N=14) | Sertraline 100mg (N=14) | Placebo (N=14)
jitteriness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
agitation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
oral surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
dry mouth (General disorders) | 0 (0) | 0 (0) | 1 (1)
drowsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes